CLINICAL TRIAL: NCT06596720
Title: Evaluating the Immediate Impact of Aerobic Exercise on Cognitive Function in Individuals Affected by Chronıc Stroke
Brief Title: Acute Effects of Aerobic Exercise on Cognitive Functions in Patients with Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emre BASKAN (Other)
Responsible Party: Sponsor-Investigator, Emre BASKAN, Associate Proffesor, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60116787-020/46559
Record Dates: First submitted 2024-08-23; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aerobic Exercise; Chronic Stroke; Cognitive Function
Keywords: aerobic exercise; chronic stroke; cognitive function
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: For cognitive assessments of the individuals, the Standardized Mini-Mental State Examination, Stroop Test, T-BAG form, Wechsler Digit Span subtest, and Letter Cancellation Test were used. The individuals with stroke in the study group underwent 30 minutes of moderate-intensity cycling on a cycle ergometer. The individuals with stroke in the control group were left in a quiet room for 30 minutes. After this period, both groups had their pulse, saturation, and blood pressure measured again, and the Stroop Test T-BAG Form, Wechsler Digit Span Tests, and Letter Cancellation Tests were repeated.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Cognitive assessments for participants in the study group were conducted using the Standardized Mini-Mental State Test, Stroop Test T-BAG Form, Wechsler Digit Span subtest, and Letter Cancellation Test. Participants underwent a thirty-minute session on a moderate-intensity bicycle ergometer. Subsequently, pulse, oxygen saturation, and blood pressure were measured, and the Stroop Test T-BAG Form, Wechsler Digit Span Tests, and Letter Cancellation Tests were repeated.
  Interventions: Other: Aerobic Exercise
- Control group (No Intervention): Cognitive assessments for participants in the control group were conducted using the Standardized Mini-Mental State Test, Stroop Test T-BAG Form, Wechsler Digit Span subtest, and Letter Cancellation Test. The control group was left in a quiet room for thirty minutes. After this period, pulse, oxygen saturation, and blood pressure were measured, and the Stroop Test T-BAG Form, Wechsler Digit Span Tests, and Letter Cancellation Tests were repeated

INTERVENTIONS:
Other: Aerobic Exercise — After the initial assessments of the individuals in the study group were completed, the exercise program was implemented. The exercise program consisted of 30 minutes of submaximal cycling using the Karvonen formula. The aerobic exercise program was structured with a 5-minute warm-up, a 5-minute cool-down, and the remaining time dedicated to the exercise phase. Since our study included only a single exercise session, a moderate-intensity training program was applied to the participants.
  Arms: Study group

SUMMARY:
The aim of this observational study is to investigate the acute effects of aerobic exercise on cognitive functions in patients with chronic stroke. The primary question addressed is:

Does aerobic exercise have an impact on cognitive functions in individuals with chronic stroke? Participants with chronic stroke were divided into two groups: those engaging in aerobic exercise and a control group. Both groups underwent cognitive function assessments at intervals of thirty minutes.

DETAILED DESCRIPTION:
WORKPLACE The study was conducted at the Department of Neurological Rehabilitation, Faculty of Physiotherapy and Rehabilitation, Pamukkale University.

PARTICIPANTS The study included 38 stroke patients admitted to Pamukkale University Hospital, aged between 25 and 80, who had a diagnosed cardiopulmonary disease or additional neurological disorders, and did not have defined psychological issues. Individuals with visual or auditory impairments were excluded from the study. Participants were informed about the study, provided with a voluntary information form to read, and written consent was obtained.

In this study, a bicycle ergometer was used considering the safety and individual capabilities of the participants. The protocol consisted of a 5-minute warm-up, 20 minutes of moderate-intensity exercise, and a 5-minute cool-down period. While most studies aim for high-intensity exercise (60-80%), this study focused on a single-session exercise training model; hence, the exercise program for the study group was set at a moderate intensity (40-50%). Participants in the study group wore a pulse oximeter and were instructed to exercise within the specified heart rate ranges. Neuropsychological tests were administered before and after the bicycle ergometer sessions. The control group underwent neuropsychological tests at thirty-minute intervals without using the bicycle ergometer.

REGISTRATION FORM The registration form collected information on demographic data, including the date of stroke onset, medical history, family history, smoking and alcohol use, dominant and affected extremities, and current comorbidities.

ASSESSMENT Participants were randomly assigned to the study or control group using a closed-envelope method. All assessments were conducted in a well-lit and quiet room. Cognitive levels were measured using the Standardized Mini-Mental State Test (SMMT). In the study group, blood pressure, pulse, and oxygen saturation were measured. Subsequently, the Stroop Test T-BAG Form, Letter Cancellation Test, and Wechsler Digit Span Test were administered. After the tests, a thirty-minute submaximal bicycle ergometer session, including a 5-minute warm-up and a 5-minute cool-down period, was conducted. Blood pressure, pulse, and oxygen saturation were measured again, and the tests were repeated. In the control group, blood pressure, pulse, and oxygen saturation were measured before administering the Stroop Test, Letter Cancellation Test, and Wechsler Digit Span Test. To avoid learning effects in the neuropsychological test battery, participants in the control group waited for approximately thirty minutes before repeating cognitive tests, and results were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Having experienced an ischemic or hemorrhagic stroke
* Having been diagnosed with a stroke at least six months prior
* Having not experienced multiple stroke episodes
* Having no communication difficulties
* Being literate

Exclusion Criteria:

* Having hearing loss
* Receiving additional treatment beyond rehabilitation
* Using a pacemaker
* Presence of cardio-pulmonary disease
* Having experienced a recent trauma
* Having additional neurological disorders aside from stroke
* Having a psychological disorder
* Having a pre-existing condition that affects cognitive level

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Stroop tests | 10 minutes
  This test is a brief measure of selective or focused attention, specifically assessing the ability to shift from one perceptual state to another and suppress response tendencies.
Wechsler Forward Digit Span, Wechsler Backward Digit Span | 10 minutes
  This test is used to assess attention and short-term memory.
CancellationTest | 5 minutes
  This test measures sustained attention, visual scanning, reaction time, and response impulsivity.

OTHER OUTCOMES:
Saturation | 5 minutes
  Oxygen saturation indicates the normal level of oxygen transported to tissues. It is a key indicator, especially for monitoring cardiopulmonary health.
Pulse values | 5 minutes
  The total number of systolic contractions of the heart per minute is referred to as the heart rate (HR), also known as the pulse.
Systolic and diastolic blood pressure | 5 minutes
  Blood pressure refers to the force exerted by blood on the inner walls of the arteries. It is one of the most fundamental indicators of a person's health. During ventricular systole, blood is ejected into the arteries, reaching its peak pressure, known as systolic pressure. During ventricular diastole, blood is drawn back, and the pressure falls to its lowest level, known as diastolic pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No